CLINICAL TRIAL: NCT02446236
Title: Phase Ib Dose Finding Study of Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib (PCI-32765) Plus Lenalidomide / Rituximab in Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Brief Title: Dose Finding Study of Ibrutinib Plus Lenalidomide / Rituximab in Relapsed or Refractory Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro 5444
Record Dates: First submitted 2015-05-06; First posted 2015-05-18 (Estimated); Results first posted 2024-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide; ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation Study (Experimental): Ibrutinib 560 mg/daily rituximab 375mg/m2 IV Day 1 Lenalidomide 10-25 mg PO days 1-21
  Interventions: Drug: Lenalidomide; Drug: Ibrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Dose escalation of lenalidomide. Patients will receive 10, 15, 20, or 25 mg PO days 1-21
  Other Names: Revlimid
Drug: Ibrutinib — 560 mg PO daily
  Other Names: Imbruvica
Drug: Rituximab — 375 mg/m2 IV Day 1
  Other Names: Rituxan

SUMMARY:
This is a dose-escalation to determine the MTD and/or RPII for combinations of ibrutinib (PCI-32765) plus lenalidomide/rituximab in patients with relapsed/refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is a relatively rare subtype (3% to 6% (Zhou, 2008) of mature B cell non-Hodgkin lymphomas (NHL), with a median age at diagnosis in mid to late 60's, a male predominance (3/1) and typically advanced stage presentation though only about 1/3 of patients are truly symptomatic at baseline (Armitage, 1998). Although significant controversies remain in the management of MCL, all would agree that the challenges associated with MCL, particularly the poor results with standard chemotherapy and frequent chemoresistance have pushed the community to be more innovative and active in clinical research. Hence the median OS has clearly improved over the last 3 decades (from 2-3y to >5y) (Goy, 2011a), thanks to deeper responses obtained with intensive regimens in younger patients (an early CR translates into clearly better outcome) and also better salvage therapies with now MCL being the only lymphoma with 4 new biologicals approved (3 in the US and 1 in EU).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Histologically or cytologically confirmed diagnosis of MCL.
* Relapsed or refractory MCL patients who have received at least one prior therapy are eligible. Patients who have previously received high-dose chemotherapy with peripheral stem cell support are eligible.
* Presence of at least one lymph node evaluable or mass measurable for response.
* Eastern Cooperative Oncology Group Performance Status greater than 2.
* Platelets > 75,000/μL and absolute neutrophils count (ANC) > 1,000/μL within 14 days of study registration (unless the treating physician deems the neutropenia is related to bone marrow involvement, then an ANC of > 750/mm 3 is allowed)
* Normal renal function defined as serum creatinine less than 2.
* Recovery from any previous treatment therapy.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Ability to understand, and willingness to sign, a written informed consent document.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anti-coagulation (patients intolerant to ASA may use low molecular weight heparin).
* Normal organ and bone marrow function parameter:

Laboratory tests Required value WBC >3000/μL* Absolute neutrophils count >1,000/μL* Platelets >75,000/μL Total bilirubin < 1.5Within normal institutional limits AST (SGOT) and ALT (SGPT) <3 x institutional upper limit of normal Creatinine or creatinine clearance <1.5 within normal institutional limits >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal (calculated by Cockcroft-Gault formula)

Exclusion Criteria:

* Concomitant use of warfarin or other Vit K antagonists
* Central nervous system (CNS) involvement by lymphoma at time of enrollment.
* Other medical conditions that would potentially interfere with patient participation in this trial.
* A second malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix (unless for other tumor type patient was treated with curative intent at least 2 years previously.)
* Known human immunodeficiency virus (HIV-1) infection or chronic hepatitis B, or C (Hep B serology positive without active infection will be eligible)
* Active, clinically serious infection > CTCAE grade 2. Patients may be eligible upon resolution of the infection.
* Major surgery or significant traumatic injury within 28 days of the first dose of study drug.
* Use of any other standard chemotherapy, radiation therapy, or experimental drug therapy for the treatment of MCL within 21 days of starting treatment or 5 half life times (whatever is shorter)
* Patients with grade 3/4 cardiac problems, as defined by the New York Heart Association (NYHA) criteria:
* History of uncontrolled or symptomatic angina
* History of uncontrolled arrhythmias
* Myocardial infarction < 6 months from study entry
* Uncontrolled or symptomatic congestive heart failure
* Ejection fraction below the institutional normal limit
* Any other cardiac condition that, in the opinion of the treatment physician, would make this protocol unreasonably hazardous for the patient
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Goy, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Ansell SM, Inwards DJ, Rowland KM Jr, Flynn PJ, Morton RF, Moore DF Jr, Kaufmann SH, Ghobrial I, Kurtin PJ, Maurer M, Allmer C, Witzig TE. Low-dose, single-agent temsirolimus for relapsed mantle cell lymphoma: a phase 2 trial in the North Central Cancer Treatment Group. Cancer. 2008 Aug 1;113(3):508-14. doi: 10.1002/cncr.23580. PMID 18543327
- [Background] Armitage JO. Management of mantle cell lymphoma. Oncology (Williston Park). 1998 Oct;12(10 Suppl 8):49-55. PMID 9830633
- [Background] Caballero D, Campo E, Lopez-Guillermo A, Martin A, Arranz-Saez R, Gine E, Lopez A, Gonzalez-Barca E, Canales MA, Gonzalez-Diaz M, Orfao A. Clinical practice guidelines for diagnosis, treatment, and follow-up of patients with mantle cell lymphoma. Recommendations from the GEL/TAMO Spanish Cooperative Group. Ann Hematol. 2013 Sep;92(9):1151-79. doi: 10.1007/s00277-013-1783-4. Epub 2013 May 29. PMID 23716187
- [Background] Corral LG, Kaplan G. Immunomodulation by thalidomide and thalidomide analogues. Ann Rheum Dis. 1999 Nov;58 Suppl 1(Suppl 1):I107-13. doi: 10.1136/ard.58.2008.i107. No abstract available. PMID 10577986
- [Background] Crane E, List A. Immunomodulatory drugs. Cancer Invest. 2005;23(7):625-34. doi: 10.1080/07357900500283101. PMID 16305990
- [Background] Davies F, Baz R. Lenalidomide mode of action: linking bench and clinical findings. Blood Rev. 2010 Nov;24 Suppl 1:S13-9. doi: 10.1016/S0268-960X(10)70004-7. PMID 21126632
- [Background] Dredge K, Horsfall R, Robinson SP, Zhang LH, Lu L, Tang Y, Shirley MA, Muller G, Schafer P, Stirling D, Dalgleish AG, Bartlett JB. Orally administered lenalidomide (CC-5013) is anti-angiogenic in vivo and inhibits endothelial cell migration and Akt phosphorylation in vitro. Microvasc Res. 2005 Jan;69(1-2):56-63. doi: 10.1016/j.mvr.2005.01.002. PMID 15797261
- [Background] Fisher RI, Bernstein SH, Kahl BS, Djulbegovic B, Robertson MJ, de Vos S, Epner E, Krishnan A, Leonard JP, Lonial S, Stadtmauer EA, O'Connor OA, Shi H, Boral AL, Goy A. Multicenter phase II study of bortezomib in patients with relapsed or refractory mantle cell lymphoma. J Clin Oncol. 2006 Oct 20;24(30):4867-74. doi: 10.1200/JCO.2006.07.9665. Epub 2006 Sep 25. PMID 17001068
- [Background] Geisler CH, Kolstad A, Laurell A, Andersen NS, Pedersen LB, Jerkeman M, Eriksson M, Nordstrom M, Kimby E, Boesen AM, Kuittinen O, Lauritzsen GF, Nilsson-Ehle H, Ralfkiaer E, Akerman M, Ehinger M, Sundstrom C, Langholm R, Delabie J, Karjalainen-Lindsberg ML, Brown P, Elonen E; Nordic Lymphoma Group. Long-term progression-free survival of mantle cell lymphoma after intensive front-line immunochemotherapy with in vivo-purged stem cell rescue: a nonrandomized phase 2 multicenter study by the Nordic Lymphoma Group. Blood. 2008 Oct 1;112(7):2687-93. doi: 10.1182/blood-2008-03-147025. Epub 2008 Jul 14. PMID 18625886
- [Background] Goy A, Sinha R, Williams ME, Kalayoglu Besisik S, Drach J, Ramchandren R, Zhang L, Cicero S, Fu T, Witzig TE. Single-agent lenalidomide in patients with mantle-cell lymphoma who relapsed or progressed after or were refractory to bortezomib: phase II MCL-001 (EMERGE) study. J Clin Oncol. 2013 Oct 10;31(29):3688-95. doi: 10.1200/JCO.2013.49.2835. Epub 2013 Sep 3. PMID 24002500
- [Background] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- [Background] Goy A, Bernstein SH, Kahl BS, Djulbegovic B, Robertson MJ, de Vos S, Epner E, Krishnan A, Leonard JP, Lonial S, Nasta S, O'Connor OA, Shi H, Boral AL, Fisher RI. Bortezomib in patients with relapsed or refractory mantle cell lymphoma: updated time-to-event analyses of the multicenter phase 2 PINNACLE study. Ann Oncol. 2009 Mar;20(3):520-5. doi: 10.1093/annonc/mdn656. Epub 2008 Dec 12. PMID 19074748
- [Background] Goy A. Are we improving the survival of patients with mantle cell lymphoma: if so, what is the explanation? Leuk Lymphoma. 2011 Oct;52(10):1828-30. doi: 10.3109/10428194.2011.604753. Epub 2011 Aug 24. No abstract available. PMID 21767240
- [Background] Goy A, Kahl B. Mantle cell lymphoma: the promise of new treatment options. Crit Rev Oncol Hematol. 2011 Oct;80(1):69-86. doi: 10.1016/j.critrevonc.2010.09.003. Epub 2010 Dec 17. PMID 21168343
- [Background] Habermann TM, Lossos IS, Justice G, Vose JM, Wiernik PH, McBride K, Wride K, Ervin-Haynes A, Takeshita K, Pietronigro D, Zeldis JB, Tuscano JM. Lenalidomide oral monotherapy produces a high response rate in patients with relapsed or refractory mantle cell lymphoma. Br J Haematol. 2009 May;145(3):344-9. doi: 10.1111/j.1365-2141.2009.07626.x. Epub 2009 Feb 24. PMID 19245430
- [Background] Hendriks RW, Yuvaraj S, Kil LP. Targeting Bruton's tyrosine kinase in B cell malignancies. Nat Rev Cancer. 2014 Apr;14(4):219-32. doi: 10.1038/nrc3702. PMID 24658273
- [Background] Herman SE, Gordon AL, Hertlein E, Ramanunni A, Zhang X, Jaglowski S, Flynn J, Jones J, Blum KA, Buggy JJ, Hamdy A, Johnson AJ, Byrd JC. Bruton tyrosine kinase represents a promising therapeutic target for treatment of chronic lymphocytic leukemia and is effectively targeted by PCI-32765. Blood. 2011 Jun 9;117(23):6287-96. doi: 10.1182/blood-2011-01-328484. Epub 2011 Mar 21. PMID 21422473
- [Background] Hernandez-Ilizaliturri FJ, Reddy N, Holkova B, Ottman E, Czuczman MS. Immunomodulatory drug CC-5013 or CC-4047 and rituximab enhance antitumor activity in a severe combined immunodeficient mouse lymphoma model. Clin Cancer Res. 2005 Aug 15;11(16):5984-92. doi: 10.1158/1078-0432.CCR-05-0577. PMID 16115943
- [Background] Hess G, Herbrecht R, Romaguera J, Verhoef G, Crump M, Gisselbrecht C, Laurell A, Offner F, Strahs A, Berkenblit A, Hanushevsky O, Clancy J, Hewes B, Moore L, Coiffier B. Phase III study to evaluate temsirolimus compared with investigator's choice therapy for the treatment of relapsed or refractory mantle cell lymphoma. J Clin Oncol. 2009 Aug 10;27(23):3822-9. doi: 10.1200/JCO.2008.20.7977. Epub 2009 Jul 6. PMID 19581539
- [Background] Hoster E, Dreyling M, Klapper W, Gisselbrecht C, van Hoof A, Kluin-Nelemans HC, Pfreundschuh M, Reiser M, Metzner B, Einsele H, Peter N, Jung W, Wormann B, Ludwig WD, Duhrsen U, Eimermacher H, Wandt H, Hasford J, Hiddemann W, Unterhalt M; German Low Grade Lymphoma Study Group (GLSG); European Mantle Cell Lymphoma Network. A new prognostic index (MIPI) for patients with advanced-stage mantle cell lymphoma. Blood. 2008 Jan 15;111(2):558-65. doi: 10.1182/blood-2007-06-095331. Epub 2007 Oct 25. PMID 17962512
- [Background] Katzenberger T, Petzoldt C, Holler S, Mader U, Kalla J, Adam P, Ott MM, Muller-Hermelink HK, Rosenwald A, Ott G. The Ki67 proliferation index is a quantitative indicator of clinical risk in mantle cell lymphoma. Blood. 2006 Apr 15;107(8):3407. doi: 10.1182/blood-2005-10-4079. No abstract available. PMID 16597597
- [Background] LaCasce AS, Vandergrift JL, Rodriguez MA, Abel GA, Crosby AL, Czuczman MS, Nademanee AP, Blayney DW, Gordon LI, Millenson M, Vanderplas A, Lepisto EM, Zelenetz AD, Niland J, Friedberg JW. Comparative outcome of initial therapy for younger patients with mantle cell lymphoma: an analysis from the NCCN NHL Database. Blood. 2012 Mar 1;119(9):2093-9. doi: 10.1182/blood-2011-07-369629. Epub 2012 Jan 10. PMID 22234679
- [Background] Leonard JP, Jung SH, Johnson J, Pitcher BN, Bartlett NL, Blum KA, Czuczman M, Giguere JK, Cheson BD. Randomized Trial of Lenalidomide Alone Versus Lenalidomide Plus Rituximab in Patients With Recurrent Follicular Lymphoma: CALGB 50401 (Alliance). J Clin Oncol. 2015 Nov 1;33(31):3635-40. doi: 10.1200/JCO.2014.59.9258. Epub 2015 Aug 24. PMID 26304886
- [Background] Lopez-Girona A, Heintel D, Zhang LH, Mendy D, Gaidarova S, Brady H, Bartlett JB, Schafer PH, Schreder M, Bolomsky A, Hilgarth B, Zojer N, Gisslinger H, Ludwig H, Daniel T, Jager U, Chopra R. Lenalidomide downregulates the cell survival factor, interferon regulatory factor-4, providing a potential mechanistic link for predicting response. Br J Haematol. 2011 Aug;154(3):325-36. doi: 10.1111/j.1365-2141.2011.08689.x. Epub 2011 Jun 24. PMID 21707574
- [Background] Lyman GH, Khorana AA, Kuderer NM, Lee AY, Arcelus JI, Balaban EP, Clarke JM, Flowers CR, Francis CW, Gates LE, Kakkar AK, Key NS, Levine MN, Liebman HA, Tempero MA, Wong SL, Prestrud AA, Falanga A; American Society of Clinical Oncology Clinical Practice. Venous thromboembolism prophylaxis and treatment in patients with cancer: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2013 Jun 10;31(17):2189-204. doi: 10.1200/JCO.2013.49.1118. Epub 2013 May 13. PMID 23669224
- [Background] Marriott JB, Clarke IA, Dredge K, Muller G, Stirling D, Dalgleish AG. Thalidomide and its analogues have distinct and opposing effects on TNF-alpha and TNFR2 during co-stimulation of both CD4(+) and CD8(+) T cells. Clin Exp Immunol. 2002 Oct;130(1):75-84. doi: 10.1046/j.1365-2249.2002.01954.x. PMID 12296856
- [Background] O'Brien SM. Update on ibrutinib. Clin Adv Hematol Oncol. 2013 Nov;11(11):735-7. No abstract available. PMID 24896547
- [Background] Ponader S, Chen SS, Buggy JJ, Balakrishnan K, Gandhi V, Wierda WG, Keating MJ, O'Brien S, Chiorazzi N, Burger JA. The Bruton tyrosine kinase inhibitor PCI-32765 thwarts chronic lymphocytic leukemia cell survival and tissue homing in vitro and in vivo. Blood. 2012 Feb 2;119(5):1182-9. doi: 10.1182/blood-2011-10-386417. Epub 2011 Dec 16. PMID 22180443
- [Background] Qian Z, Zhang L, Cai Z, Sun L, Wang H, Yi Q, Wang M. Lenalidomide synergizes with dexamethasone to induce growth arrest and apoptosis of mantle cell lymphoma cells in vitro and in vivo. Leuk Res. 2011 Mar;35(3):380-6. doi: 10.1016/j.leukres.2010.09.027. Epub 2010 Nov 2. PMID 21047686
- [Background] Ramsay AG, Clear AJ, Kelly G, Fatah R, Matthews J, Macdougall F, Lister TA, Lee AM, Calaminici M, Gribben JG. Follicular lymphoma cells induce T-cell immunologic synapse dysfunction that can be repaired with lenalidomide: implications for the tumor microenvironment and immunotherapy. Blood. 2009 Nov 19;114(21):4713-20. doi: 10.1182/blood-2009-04-217687. Epub 2009 Sep 28. PMID 19786615
- [Background] Rickert RC. New insights into pre-BCR and BCR signalling with relevance to B cell malignancies. Nat Rev Immunol. 2013 Aug;13(8):578-91. doi: 10.1038/nri3487. PMID 23883968
- [Background] Romaguera JE, Fayad L, Rodriguez MA, Broglio KR, Hagemeister FB, Pro B, McLaughlin P, Younes A, Samaniego F, Goy A, Sarris AH, Dang NH, Wang M, Beasley V, Medeiros LJ, Katz RL, Gagneja H, Samuels BI, Smith TL, Cabanillas FF. High rate of durable remissions after treatment of newly diagnosed aggressive mantle-cell lymphoma with rituximab plus hyper-CVAD alternating with rituximab plus high-dose methotrexate and cytarabine. J Clin Oncol. 2005 Oct 1;23(28):7013-23. doi: 10.1200/JCO.2005.01.1825. Epub 2005 Sep 6. PMID 16145068
- [Background] Rosenwald A, Wright G, Wiestner A, Chan WC, Connors JM, Campo E, Gascoyne RD, Grogan TM, Muller-Hermelink HK, Smeland EB, Chiorazzi M, Giltnane JM, Hurt EM, Zhao H, Averett L, Henrickson S, Yang L, Powell J, Wilson WH, Jaffe ES, Simon R, Klausner RD, Montserrat E, Bosch F, Greiner TC, Weisenburger DD, Sanger WG, Dave BJ, Lynch JC, Vose J, Armitage JO, Fisher RI, Miller TP, LeBlanc M, Ott G, Kvaloy S, Holte H, Delabie J, Staudt LM. The proliferation gene expression signature is a quantitative integrator of oncogenic events that predicts survival in mantle cell lymphoma. Cancer Cell. 2003 Feb;3(2):185-97. doi: 10.1016/s1535-6108(03)00028-x. PMID 12620412
- [Background] Rummel MJ, Niederle N, Maschmeyer G, Banat GA, von Grunhagen U, Losem C, Kofahl-Krause D, Heil G, Welslau M, Balser C, Kaiser U, Weidmann E, Durk H, Ballo H, Stauch M, Roller F, Barth J, Hoelzer D, Hinke A, Brugger W; Study group indolent Lymphomas (StiL). Bendamustine plus rituximab versus CHOP plus rituximab as first-line treatment for patients with indolent and mantle-cell lymphomas: an open-label, multicentre, randomised, phase 3 non-inferiority trial. Lancet. 2013 Apr 6;381(9873):1203-10. doi: 10.1016/S0140-6736(12)61763-2. Epub 2013 Feb 20. PMID 23433739
- [Background] Satterthwaite AB, Willis F, Kanchanastit P, Fruman D, Cantley LC, Helgason CD, Humphries RK, Lowell CA, Simon M, Leitges M, Tarakhovsky A, Tedder TF, Lesche R, Wu H, Witte ON. A sensitized genetic system for the analysis of murine B lymphocyte signal transduction pathways dependent on Bruton's tyrosine kinase. Proc Natl Acad Sci U S A. 2000 Jun 6;97(12):6687-92. doi: 10.1073/pnas.110146697. PMID 10829070
- [Background] Schafer PH, Gandhi AK, Loveland MA, Chen RS, Man HW, Schnetkamp PP, Wolbring G, Govinda S, Corral LG, Payvandi F, Muller GW, Stirling DI. Enhancement of cytokine production and AP-1 transcriptional activity in T cells by thalidomide-related immunomodulatory drugs. J Pharmacol Exp Ther. 2003 Jun;305(3):1222-32. doi: 10.1124/jpet.102.048496. Epub 2003 Mar 20. PMID 12649301
- [Background] Shaffer AL, Rosenwald A, Staudt LM. Lymphoid malignancies: the dark side of B-cell differentiation. Nat Rev Immunol. 2002 Dec;2(12):920-32. doi: 10.1038/nri953. PMID 12461565
- [Background] Tam CS, Khouri IF. Autologous and allogeneic stem cell transplantation: rising therapeutic promise for mantle cell lymphoma. Leuk Lymphoma. 2009 Aug;50(8):1239-48. doi: 10.1080/10428190903026518. PMID 19562639
- [Background] Vegliante MC, Palomero J, Perez-Galan P, Roue G, Castellano G, Navarro A, Clot G, Moros A, Suarez-Cisneros H, Bea S, Hernandez L, Enjuanes A, Jares P, Villamor N, Colomer D, Martin-Subero JI, Campo E, Amador V. SOX11 regulates PAX5 expression and blocks terminal B-cell differentiation in aggressive mantle cell lymphoma. Blood. 2013 Mar 21;121(12):2175-85. doi: 10.1182/blood-2012-06-438937. Epub 2013 Jan 15. PMID 23321250
- [Background] Verhelle D, Corral LG, Wong K, Mueller JH, Moutouh-de Parseval L, Jensen-Pergakes K, Schafer PH, Chen R, Glezer E, Ferguson GD, Lopez-Girona A, Muller GW, Brady HA, Chan KW. Lenalidomide and CC-4047 inhibit the proliferation of malignant B cells while expanding normal CD34+ progenitor cells. Cancer Res. 2007 Jan 15;67(2):746-55. doi: 10.1158/0008-5472.CAN-06-2317. PMID 17234786
- [Background] Vose JM. Mantle cell lymphoma: 2012 update on diagnosis, risk-stratification, and clinical management. Am J Hematol. 2012 Jun;87(6):604-9. doi: 10.1002/ajh.23176. PMID 22615102
- [Background] Wang ML, Rule S, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Li L, Zhang L, Newberry K, Ou Z, Cheng N, Fang B, McGreivy J, Clow F, Buggy JJ, Chang BY, Beaupre DM, Kunkel LA, Blum KA. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med. 2013 Aug 8;369(6):507-16. doi: 10.1056/NEJMoa1306220. Epub 2013 Jun 19. PMID 23782157
- [Background] Wang M, Fowler N, Wagner-Bartak N, Feng L, Romaguera J, Neelapu SS, Hagemeister F, Fanale M, Oki Y, Pro B, Shah J, Thomas S, Younes A, Hosing C, Zhang L, Newberry KJ, Desai M, Cheng N, Badillo M, Bejarano M, Chen Y, Young KH, Champlin R, Kwak L, Fayad L. Oral lenalidomide with rituximab in relapsed or refractory diffuse large cell, follicular and transformed lymphoma: a phase II clinical trial. Leukemia. 2013 Sep;27(9):1902-9. doi: 10.1038/leu.2013.95. Epub 2013 Apr 2. PMID 23545991
- [Background] Wiernik PH, Lossos IS, Tuscano JM, Justice G, Vose JM, Cole CE, Lam W, McBride K, Wride K, Pietronigro D, Takeshita K, Ervin-Haynes A, Zeldis JB, Habermann TM. Lenalidomide monotherapy in relapsed or refractory aggressive non-Hodgkin's lymphoma. J Clin Oncol. 2008 Oct 20;26(30):4952-7. doi: 10.1200/JCO.2007.15.3429. Epub 2008 Jul 7. PMID 18606983
- [Background] Witzig TE, Vose JM, Zinzani PL, Reeder CB, Buckstein R, Polikoff JA, Bouabdallah R, Haioun C, Tilly H, Guo P, Pietronigro D, Ervin-Haynes AL, Czuczman MS. An international phase II trial of single-agent lenalidomide for relapsed or refractory aggressive B-cell non-Hodgkin's lymphoma. Ann Oncol. 2011 Jul;22(7):1622-1627. doi: 10.1093/annonc/mdq626. Epub 2011 Jan 12. PMID 21228334
- [Background] Witzig TE, Geyer SM, Ghobrial I, Inwards DJ, Fonseca R, Kurtin P, Ansell SM, Luyun R, Flynn PJ, Morton RF, Dakhil SR, Gross H, Kaufmann SH. Phase II trial of single-agent temsirolimus (CCI-779) for relapsed mantle cell lymphoma. J Clin Oncol. 2005 Aug 10;23(23):5347-56. doi: 10.1200/JCO.2005.13.466. Epub 2005 Jun 27. PMID 15983389
- [Background] Wodarz D, Garg N, Komarova NL, Benjamini O, Keating MJ, Wierda WG, Kantarjian H, James D, O'Brien S, Burger JA. Kinetics of CLL cells in tissues and blood during therapy with the BTK inhibitor ibrutinib. Blood. 2014 Jun 26;123(26):4132-5. doi: 10.1182/blood-2014-02-554220. Epub 2014 May 14. PMID 24829205
- [Background] Woyach JA, Smucker K, Smith LL, Lozanski A, Zhong Y, Ruppert AS, Lucas D, Williams K, Zhao W, Rassenti L, Ghia E, Kipps TJ, Mantel R, Jones J, Flynn J, Maddocks K, O'Brien S, Furman RR, James DF, Clow F, Lozanski G, Johnson AJ, Byrd JC. Prolonged lymphocytosis during ibrutinib therapy is associated with distinct molecular characteristics and does not indicate a suboptimal response to therapy. Blood. 2014 Mar 20;123(12):1810-7. doi: 10.1182/blood-2013-09-527853. Epub 2014 Jan 10. PMID 24415539
- [Background] Wu A, Scheffler MR. Multi-dose phamacokinetics and safety of CC-5013 in 15 multiple myeloma patients. J Clin Oncol.;22:141s, 2004
- [Background] Wu L, Adams M, Carter T, Chen R, Muller G, Stirling D, Schafer P, Bartlett JB. lenalidomide enhances natural killer cell and monocyte-mediated antibody-dependent cellular cytotoxicity of rituximab-treated CD20+ tumor cells. Clin Cancer Res. 2008 Jul 15;14(14):4650-7. doi: 10.1158/1078-0432.CCR-07-4405. PMID 18628480
- [Background] Zhang L, Qian Z, Cai Z, Sun L, Wang H, Bartlett JB, Yi Q, Wang M. Synergistic antitumor effects of lenalidomide and rituximab on mantle cell lymphoma in vitro and in vivo. Am J Hematol. 2009 Sep;84(9):553-9. doi: 10.1002/ajh.21468. PMID 19565649
- [Background] Zhou X, Teegala S, Huen A, Ji Y, Fayad L, Hagemeister FB, Gladish G, Vadhan-Raj S. Incidence and risk factors of venous thromboembolic events in lymphoma. Am J Med. 2010 Oct;123(10):935-41. doi: 10.1016/j.amjmed.2010.05.021. PMID 20920696
- [Background] Zhou Y, Wang H, Fang W, Romaguer JE, Zhang Y, Delasalle KB, Kwak L, Yi Q, Du XL, Wang M. Incidence trends of mantle cell lymphoma in the United States between 1992 and 2004. Cancer. 2008 Aug 15;113(4):791-8. doi: 10.1002/cncr.23608. PMID 18615506
- [Background] Zhu D, Corral LG, Fleming YW, Stein B. Immunomodulatory drugs Revlimid (lenalidomide) and CC-4047 induce apoptosis of both hematological and solid tumor cells through NK cell activation. Cancer Immunol Immunother. 2008 Dec;57(12):1849-59. doi: 10.1007/s00262-008-0512-7. Epub 2008 Apr 8. PMID 18392823
- [Background] Zinzani PL, Vose JM, Czuczman MS, Reeder CB, Haioun C, Polikoff J, Tilly H, Zhang L, Prandi K, Li J, Witzig TE. Long-term follow-up of lenalidomide in relapsed/refractory mantle cell lymphoma: subset analysis of the NHL-003 study. Ann Oncol. 2013 Nov;24(11):2892-7. doi: 10.1093/annonc/mdt366. Epub 2013 Sep 12. PMID 24030098

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Dose Level 1: Ibrutinib 560 mg/daily rituximab 375mg/m2 IV Day 1 Lenalidomide 15mg PO days 1-21
- Phase I - Dose Level 2; Phase II Expansion: Ibrutinib 560 mg/daily rituximab 375mg/m2 IV Day 1 Lenalidomide 20 mg PO days 1-21
Period: Overall Study
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase II Expansion
Started | 5 | 3 | 19
Completed | 4 | 3 | 17
Not Completed | 1 | 0 | 2
Not completed — Screen Failure | 1 | 0 | 1
Not completed — Actively Receiving Therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase II Expansion | Total
Number analyzed (Participants) | 4 | 3 | 18 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 8 | 10
  >=65 years | 3 | 2 | 10 | 15
Age, Continuous [Median (Full Range); unit: Years] | 69.5 [58 to 70] | 71 [52 to 79] | 65.5 [47 to 82] | 67 [47 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 5 | 6
  Male | 3 | 3 | 13 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 2 | 16 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 18 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 18 | 25

OUTCOME MEASURES:

1. Primary Outcome: Determine the MTD (Measured in mg) Based on the Number of Patients With Adverse Events
Description: Define maximum tolerated dose (MTD) and /or recommended phase II dose for the combinations of Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib (PCI-32765) plus lenalidomide / rituximab in relapsed or refractory MCL by assessing the incidence of dose limiting toxicities (DLTs) in cycle 1 through an assessment of adverse events
Time Frame: 28 Days
Population: Phase I Cohorts
Measure: Number; unit: mg
Arm/Group | Dose Escalation Study
Number analyzed (Participants) | 7
mg | 20

2. Secondary Outcome: Assess Safety Profile Through Review of Adverse Events
Description: Assess safety and tolerability of the combinations through the review of adverse events. Patients will remain on treatment until disease progression or unacceptable toxicity. There is no predetermined length of treatment.
Time Frame: Through 28 Days After Discontinuation of Study Drug
Reporting Status: Not Posted

3. Secondary Outcome: Assess Radiologic Progression-Free Survival
Description: Assess preliminary anti-tumor activity of the combinations by radiological progression-free survival. Patients will remain on treatment until disease progression or unacceptable toxicity. There is no predetermined length of treatment.
Time Frame: Response is evaluated after 2, 4 and 6 cycles, after initiation of treatment and later every 3 cycles until disease progression or patient taken off study
Reporting Status: Not Posted

4. Secondary Outcome: Assess Radiologic Response Rate
Description: Assess preliminary anti-tumor activity of the combinations by radiological response rate. Patients will remain on treatment until disease progression or unacceptable toxicity. There is no predetermined length of treatment.
Time Frame: as for outcome 3
Reporting Status: Not Posted

5. Secondary Outcome: Assess Drug-drug Interaction of Combination Therapy
Description: Investigate potential drug-drug interaction between Ibrutinib (PCI-32765) plus lenalidomide / rituximab. Patients will remain on treatment until disease progression or unacceptable toxicity. There is no predetermined length of treatment.
Time Frame: Through 28 Days After Discontinuation of Study Drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase II Expansion
All-Cause Mortality (participants affected / at risk) | 1/4 | 2/3 | 2/18
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/3 | 11/18
Other Adverse Events (participants affected / at risk) | 2/4 | 2/3 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1 (N=4) | Phase I - Dose Level 2 (N=3) | Phase II Expansion (N=18)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (Investigations) | 0 (0) | 0 (0) | 3 (3)
GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Preseptal Orbital Cellulitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Psychiatric Decompensation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic Sacrolitiis and Osteomyelitis with Numerous Abscesses (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1 (N=4) | Phase I - Dose Level 2 (N=3) | Phase II Expansion (N=18)
Arrythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes